CLINICAL TRIAL: NCT04231409
Title: Study to Demonstrate the Value of Fast-Acting Subperception (FAST) Using the Spectra WaveWriter™ Spinal Cord Stimulator System in the Treatment of Chronic Pain (COMBO Study)
Brief Title: Fast-Acting Subperception Study (FAST)
Acronym: FAST
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study follow-up activities affected by COVID-19
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 92285183
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Results first posted 2022-01-24 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- WaveWriter Settings (Active Comparator): WaveWriter Programming
  Interventions: Device: Boston Scientific Spectra WaveWriter SCS System
- Conventional Settings (Active Comparator): Conventional Programming
  Interventions: Device: Boston Scientific Spectra WaveWriter SCS System

INTERVENTIONS:
Device: Boston Scientific Spectra WaveWriter SCS System — The Spectra WaveWriter Spinal Cord Stimulator (SCS) System is indicated as an aid in the management of chronic intractable pain of the trunk and/or limbs, including unilateral or bilateral pain associated with the following: failed back surgery syndrome, Complex Regional Pain Syndrome (CRPS) Types I and II, intractable low back pain and leg pain.

SUMMARY:
Study to Demonstrate the Value of Fast-Acting Subperception (FAST) using the Spectra WaveWriter™ Spinal Cord Stimulator System in the Treatment of Chronic Pain

ELIGIBILITY:
Key Inclusion Criteria:

* Chronic pain of the trunk and/or limbs for at least 6 months with back pain greater or equal to leg pain.
* 22 years of age or older at time of enrollment
* Able to independently read and complete all questionnaires and assessments provided in English
* Signed a valid, IRB-approved informed consent form (ICF) provided in English

Key Exclusion Criteria:

* Any pain-related diagnosis or medical/psychological condition that, in the clinician's best judgment, might confound reporting of study outcomes
* Significant cognitive impairment that, in the opinion of the Investigator, would reasonably be expected to impair the study candidate's ability to participate in the study
* Breast-feeding or planning to get pregnant during the course of the study or not using adequate contraception
* Participating, or intends to participate, in another clinical trial that may influence the data that will be collected for this study

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-11-26 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Wallace, Principal Investigator — University of California, San Diego
Locations (6):
- United States (6):
  - Center for Pain and Supportive Care, Phoenix, Arizona
  - Willis-Knighton River Cities Clinical Research Center, Shreveport, Louisiana
  - The Center for Clinical Research, LLC, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Pacific Sports and Spine, LLC, Eugene, Oregon
  - Precision Spine Care, Tyler, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: After subjects were enrolled, they were evaluated per study eligibility criteria. Only those who met all criteria proceeded to receive implant and randomized in the study (as applicable).
Period: Overall Study
Arm/Group | WaveWriter Settings | Conventional Settings
Started | 5 | 4
Completed | 0 | 0
Not Completed | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | WaveWriter Settings | Conventional Settings | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (16.5) | 57.3 (7.3) | 58.3 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 3 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Overall Pain Score [Mean (Standard Deviation); unit: units on a scale] — Overall Pain Score measured on a scale of 0 - 10 where 0 is no pain and 10 is worse pain possible.
  units on a scale | 7.6 (0.9) | 7.3 (1.0) | 7.4 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: Overall Pain Responder Rate
Description: Proportion of subjects with 50% or greater reduction from Baseline Visit in average overall pain intensity at 3 months post-randomization
Time Frame: 3 months post-randomization
Population: Data not collected and hence not available due to termination of the study (Follow-up activities affected by COVID-19)
Arm/Group | WaveWriter Settings | Conventional Settings
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events up to end of randomized phase (3 months)
Arm/Group | WaveWriter Settings | Conventional Settings
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 2/5 | 0/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | WaveWriter Settings (N=5) | Conventional Settings (N=4)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Shock (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-31): https://cdn.clinicaltrials.gov/large-docs/09/NCT04231409/Prot_SAP_002.pdf